CLINICAL TRIAL: NCT06531499
Title: A Phase I, Open-label, Multi-center Study of Radiation Dosimetry, Safety, and Tolerability of Extended Lutetium (177Lu) Vipivotide Tetraxetan Treatment in Chemo-naïve Adults With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Radiation Dosimetry, Safety, and Tolerability of Extended Lutetium (177Lu) Vipivotide Tetraxetan Treatment in Chemo-naïve Adults With Metastatic Castration-resistant Prostate Cancer: RADIOpharmaceutical DOSimetry Evaluation (RADIODOSE) Study
Acronym: RADIODOSE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617A12101; 2024-512338-13 (EudraCT Number)
Record Dates: First submitted 2024-06-18; First posted 2024-08-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Phase 1; RADIODOSE; AAA617; metastatic castration-resistant prostate cancer; radiation dosimetry; mCRPC; Prostate-specific membrane antigen (PSMA); Dosimetry; [68Ga]Ga-PSMA-11; gallium (68Ga) gozetotide; [177Lu]Lu-PSMA-617; lutetium (177Lu) vipivotide tetraxetan; Radioligand Imaging (RLI); Radioligand Therapy (RLT)
MeSH Terms: interventions — Lutetium; Lutetium-177; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a treatment arm based on their PSMA expressed target per PET images (based on central read).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AAA617 (Experimental): All participants will receive the investigational product AAA617 (7.4 GBq ±10%).
  Interventions: Drug: AAA617; Drug: Gonadotropin-releasing hormone (GnRH) analogues; Drug: Gonadotropin-releasing hormone (GnRH) antagonists

INTERVENTIONS:
Drug: AAA617 — [177Lu]Lu-PSMA-617 will be administered as an intravenous infusion at a dose of 7.4 GBq (200mCi) (+/- 10%), every 6 weeks for up to 12 cycles.
  Other Names: Lutetium (177Lu) vipivotide tetraxetan, [177Lu]Lu-PSMA-617
Drug: Gonadotropin-releasing hormone (GnRH) analogues — Anatomical Therapeutic Chemical [ATC] code L02AE
Drug: Gonadotropin-releasing hormone (GnRH) antagonists — Degarelix, Relugolix

SUMMARY:
The purpose of the study is to assess and evaluate dosimetry, safety, and tolerability following administration of up to 12 cycles of (177Lu) vipivotide tetraxetan (also referred to as [177Lu]Lu-PSMA-617 or 177Lu-PSMA-617 and hereafter identified as AAA617) in taxane-naïve adult participants with PSMA-positive mCRPC who progressed on a prior ARPI treatment with normal renal function or mild renal impairment (eGFR ≥ 60ml/min).

DETAILED DESCRIPTION:
The study includes screening period, treatment period, and a post-treatment follow-up period.

Screening Period: Approximately 106 participants will be enrolled to receive up to12 consecutive cycles of AAA617. Potential participants will be assessed for eligibility by verifying their baseline PSMA PET scan for mandatory confirmation of PSMA positivity prior to first cycle by local review.

Treatment Period: Eligible participants will be treated with up to 12 cycles of 7.4 GBq AAA617 intravenously every 6 weeks, until radiographic progression, toxicity leading to treatment discontinuation, death, loss to follow-up, or withdrawal of consent, whichever occurs first. During treatment period, all participants who complete the initial 6 cycles of AAA617 treatment will undergo an additional PSMA-PET scan after Cycle 6 to re-assess PSMA expression level and to reassess eligibility of participants to receive additional AAA617 treatment cycles.

Post-Treatment Follow-Up: All participants will undergo a PSMA-PET scan at end of treatment (EOT). The post-treatment follow-up period will consist of EOT; 42-days safety; EOT RLI; safety, survival and rPFS follow-up visits.

The planned duration of treatment period is up to 74 weeks with treatment given every 6 weeks. Participants may be discontinued from treatment earlier due to unacceptable toxicity or disease progression, and/or at the discretion of the Investigator or the participant.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Participants must be adults ≥ 18 years of age.
* Participants must have an ECOG performance status ≤ 1.
* Participants must have histological confirmation of adenocarcinoma of the prostate.
* Participants must be PSMA-positive per 68Ga-PSMA PET/CT scans at baseline
* Participants must have a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L) either by pharmaceutical or surgical methods.
* Participants must have progressed only once on prior second generation ARPIs
* Documented progressive mCRPC
* Participants must have ≥ 1 metastatic lesion by conventional imaging that is present on screening/baseline CT, MRI, or bone scan
* Renal: eGFR ≥ 60 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Participants must have recovered to ≤ Grade 2 from all clinically significant toxicities related to prior therapies except alopecia.

Key exclusion Criteria:

* Previous treatment with any of the following within 6 months of study enrollment: Strontium 89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation
* Any previous radioligand therapy.
* Prior treatment with cytotoxic chemotherapy for metastatic castration-resistant or metastatic hormone-sensitive prostate cancer (mHSPC) (e.g., taxanes, platinum, estramustine, vincristine, methotrexate, etc.), immunotherapy or biological therapy [including monoclonal antibodies]. [Note: Taxane exposure (maximum 6 cycles) in the adjuvant or neoadjuvant setting is allowed if 12 months have elapsed since completion of this adjuvant or neoadjuvant therapy. Prior treatment with sipuleucel-T is allowed].
* Concurrent therapies: cytotoxic chemotherapy, immunotherapy, radioligand therapy, PARP inhibitor, biological, or investigational therapy
* History of myocardial infarction (MI), angina pectoris, or coronary artery bypass graft (CABG) within 6 months prior to ICF signature and/or clinically active significant cardiac disease
* Concurrent serious acute or chronic nephropathy and/or moderate to severe renal impairment as determined by the principal investigator.
* Diagnosed with other active malignancies that are expected to alter life expectancy or may interfere with disease assessment
* Sexually active males unwilling to use a condom during intercourse while taking study treatment and for 14 weeks after stopping study treatment.
* Concurrent urinary outflow obstruction or unmanageable urinary incontinence
* History of somatic or psychiatric disease/condition that may interfere with the aims and assessments of the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 106 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2028-11-24 (Estimated); Study Completion 2028-11-24 (Estimated)

PRIMARY OUTCOMES:
Time activity curves (TACs) and absorbed radiation dose of AAA617 in organs | From Cycle 1 to Cycle 12; cycle = 42 days
  Time activity curve (TAC) will be generated from the amount radioactivity in one given tissue. Time integrated activity coefficient and absorbed dose will be calculated
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | For up to 12 cycles in taxane-naive participants with progressive PSMA-positive mCRPC with nrmal kidney function or mild renal impairment; cycle = 42 days
  The distribution of adverse events for Radioligand Therapy (RLT) will be done via the analysis of frequencies for Adverse Event (AEs) and Serious Adverse Event (SAEs) through the monitoring of relevant clinical and laboratory safety parameters.
  Adverse event monitoring should be continued for at least 42 days following the end of treatment (EOT) visit.
  Participants receiving the study treatment will continue to be followed for safety every 12 weeks during the long-term follow-up for selected adverse events
Percentage of participants with AAA617 dose reductions, interruptions and discontinuations | Up to 42 (+7) days after last AAA617 dose administration (Safety Follow-up)
  The assessment of tolerability will be based on the frequency of participants with dose interruptions, reductions, and study treatment discontinuations. Dose reduction will be based on the worst toxicity demonstrated at the last dose.

SECONDARY OUTCOMES:
Time activity curves (TACs) and absorbed radiation dose AAA617 in tumors | For up to 12 cycles; cycle = 42 days
  Time activity curves (TACs) will be generated from the amount of radioactivity in one given tissue at a given moment. TACs will be fitted to mono- and bi-exponential curves. Time integrated activity coefficient and absorbed dose will be calculated.
Pharmacokinetic ( PK) concentration of AAA617 in blood over time | Cycle 1, Cycle 4, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11 and Cycle 12, cycle = 42 days
  PK concentrations will be listed by patient and visit/sampling time point. The descriptive summary statistics will be provided by visit/sampling time point.
Pharmacokinetic (PK) parameter Cmax of AAA617 from blood radioactivity data | Cycle 1, Cycle 4, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11 and Cycle 12; cycle = 42 days
  Derived PK parameter, Cmax will be listed by patient and visit. The descriptive summary statistics will be provided by visit.
  Cmax is the maximum drug concentration after dosing.
PK parameter Tmax of AAA617 from blood radioactivity data | Cycle 1, Cycle 4, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11 and Cycle 12; cycle = 42 days
  Derived PK parameter Tmax, will be listed by patient and visit. The descriptive summary statistics will be provided by visit.
  Tmax is the time to reach the maximum concentration.
PK parameter AUC of AAA617 from blood radioactivity data | Cycle 1, Cycle 4, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11 and Cycle 12; cycle = 42 days
  Derived PK parameter AUC will be listed by patient and visit. The descriptive summary statistics will be provided by visit.
  AUC: Area under the concentration-time curve.
PK parameter CL of AAA617 from blood radioactivity data | Cycle 1, Cycle 4, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11 and Cycle 12; cycle = 42 days
  Derived PK parameter CL will be listed by patient and visit. The descriptive summary statistics will be provided by visit.
  Clearance (CL): Rate at which the body eliminates the drug.
PK parameter VZ of AAA617 from blood radioactivity data | Cycle 1, Cycle 4, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11 and Cycle 12; cycle = 42 days
  Derived PK parameter Vz will be listed by patient and visit. The descriptive summary statistics will be provided by visit.
  Vz: volume of distribution during the terminal phase (Vz).
PK parameter terminal T1/2 of AAA617 from blood radioactivity data | Cycle 1, Cycle 4, Cycle 6, Cycle 7, Cycle 8, Cycle 9, Cycle 10, Cycle 11, and Cycle 12; cycle = 42 days
  Derived PK parameter terminal T1/2 will be listed by patient and visit. The descriptive summary statistics will be provided by visit.
  T1/2: Terminal half life.
Overall response rate (ORR) | From first patient first visit (FPFV) to end of study, until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 58 months
  ORR is defined as the proportion of participants with BOR of confirmed CR or PR per investigator assessment and according to Prostate Cancer Working Group 3 (PCWG3) modified-RECIST v1.1.
Disease Control rate (DCR) | From first patient first visit (FPFV) to end of study, until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 58 months
  DCR is defined as the percentage of CR, PR, stable disease or non-CR/non-progressive disease (PD) per investigator assessment and according to PCWG3 modified-RECIST v1.1 assessment in soft tissue, lymph node, and visceral lesions.
Duration of response (DOR) | From first patient first visit (FPFV) to end of study, until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 58 months
  DOR is defined as the duration of time between the date of the first documented BOR (CR or PR) per investigator assessment according to PCWG3 modified-RECIST v1.1 and the date of first documented progression or death due to any cause.
Radiographic Progressive free survival (rPFS) | From first patient first visit (FPFV) to end of study, until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to approximately 58 months
  rPFS defined as the time from the date of first dose of study treatment to the date of the first documented radiographic disease progression as assessed by investigator and PCWG3 modified-RECIST v1.1 criteria or death due to any cause, whichever occurs first.
Prostate specific antigen (PSA) response | Baseline, (Cycle (C), Day (D)) C1D1, C2D1, C3D1, C4D1, C5D1, C6D1, C6D42, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1, End Of Treatment (EOT), 6 weeks after EOT, every 12 weeks after EOT up to 12 months; each cycle = 42 days
  PSA response is defined as percentage of participants who achieve any decrease from baseline that is confirmed by a second PSA measurement ≥4 weeks. Participants with any decrease in PSA will also be summarized by visit.
Overall survival (OS) | Cycle 1 to death event, approx. 5 years, (cycle = 42 days)
  Overall survival is defined as the time from the first dose of study treatment to death due to any cause.
Duration of exposure to AAA617 and dose intensity | during treatment period (74 weeks)
  Duration of exposure:
  Dose intensity is computed as the ratio of actual cumulative dose received and actual duration of exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- United States (5):
  - University of California LA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Wash U School of Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
- Germany (7):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Wuppertal, North Rhine-Westphalia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Rostock
- Novartis Investigative Site, Nijmegen, Gelderland, Netherlands
- Spain (3):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Barcelona
- Switzerland (2):
  - Novartis Investigative Site, Bellinzona
  - Novartis Investigative Site, Bern
- United Kingdom (3):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Glasgow

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.